CLINICAL TRIAL: NCT01802788
Title: International Long-term Follow-up Study of Patients Implanted With a Portico™ Valve
Brief Title: 5 Year Observation of Patients With PORTICO Valves
Acronym: PORTICO-1
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CV-12-054-EU-PV
Record Dates: First submitted 2013-02-21; First posted 2013-03-01 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Stenosis; CV-12-054-EU-PV; Heart Valve Prosthesis; Trans Catheter Aortic Valve Replacement; TAVR; Trans Catheter Aortic Valve Implant; TAVI
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort A: Patients implanted with a Portico valve after CE mark
  Interventions: Device: St Jude Medical Portico replacement aortic valve; Procedure: Transcatheter Aortic Valve Implant
- Cohort B: Patients implanted in previous SJM-sponsored premarket studies
  Interventions: Device: St Jude Medical Portico replacement aortic valve; Procedure: Transcatheter Aortic Valve Implant

INTERVENTIONS:
Device: St Jude Medical Portico replacement aortic valve
Procedure: Transcatheter Aortic Valve Implant
  Other Names: TAVI; Transcatheter Aortic Valve Replacement; TAVR

SUMMARY:
The purpose of this clinical investigation is to further assess the performance and safety profile of the commercially-available Portico™ TAVI System in patients with severe symptomatic aortic stenosis.

DETAILED DESCRIPTION:
This is an international multicenter, prospective, non-randomized clinical investigation without concurrent or matched control, designed to assess the mid-term safety and performance of the Portico valve in patients with severe symptomatic aortic stenosis whom are high risk for surgical valve replacement. The primary endpoint is 1 year all-cause mortality. In addition, the performance and safety profile of the Portico valve will be further evaluated at 30 days, 1 year, and annually through 5 years post-implant.

The investigation will be conducted at approximately 65 centers in approximately 15 countries in Europe, Middle-East, Africa, Canada, Australia and New Zealand.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed the Patient Informed Consent prior to participating in the clinical investigation.
* Patient has been referred for a Portico Valve implant as per Heart Team decision or patient has received a Portico Valve as per participation in an SJM sponsored regulatory or first-in-human trial.
* Patient has senile degenerative aortic valve stenosis confirmed by echocardiographically derived criteria*:

  * An initial aortic valve area (AVA) of less than or equal to (≤) 1.0 cm2 (or indexed EOA less than or equal to (≤) 0.6 cm2/m2) AND
  * A mean gradient greater than (>)40 mmHg or jet velocity greater than (>)4.0 m/s or Doppler Velocity Index less than (<)0.25. If the mean gradient is <40 mmHg and left ventricular ejection fraction (LVEF) <55%, then the site may as well perform a dobutamine stress echo to see if the mean gradient increases to >40 mmHg." (Baseline measurement taken by echo within 6 months of index procedure.)
* Patient has a life expectancy more than (>) 12 months.

For patients enrolled in a French site:

* Patient is at high risk for surgery as demonstrated by a Logistic EuroSCORE equal or more than (≥) 20 and/or a Society of Thoracic Surgeon (STS) mortality risk score of more than (>) 10% and/or by clinical judgment of the Heart Team based on the individual risk profile (comorbidities).

  * Not applicable for a patient who has received a Portico Valve as per participation in an SJM sponsored Regulatory or First-In-Human trial.

Exclusion Criteria:

* Any case in which the Portico Valve would not be indicated for the patient as per current instructions for use (i.e any "off-label" use).
* Patient has any other aortic valve than tricuspid one.
* Patient has a prosthetic valve or ring in the aortic position.
* Patient needs a concomitant structural heart procedure..
* Patient needs the usage of an embolic protection device.
* Patient is unwilling or unable to comply with all clinical investigation-required follow-up evaluations.
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises of Cohort A and Cohort B with severe symptomatic aortic stenosis (AS).
  Cohort A: Patients enrolled directly into the Portico I study.
  Cohort B: Patients implanted in previous SJM-sponsored regulatory (pre-market) investigations and first-in-human trials whom consent for ongoing follow-up in the Portico I study after the completion of their participation in the initial study.
Sampling Method: Non-Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2013-04-16 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Maisano, MD, Principal Investigator — San Raffaele Hospital; Stephen Worthley, Principal Investigator — St Andrews Hospital; Josep Rodes-Cabau, Principal Investigator — Institut de Cardiologie de Quebec (Hospital Laval)
Locations (60):
- Australia (10):
  - Royal Adelaide Hospital, Adelaide
  - St Andrews Hospital, Adelaide
  - Heart Care Partners-Wesley Hospital, Auchenflower
  - The Prince Charles Hospital, Chermside
  - Royal North Shore hospital, Leonards Hill
  - The Alfred Hospital, Melbourne
  - Royal Melbourne Hospital - City Campus, Parkville
  - Fiona Stanley Hospital, Perth
  - North Shore Private Hospital, St Leonards
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (3):
  - AZ Middelheim, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHR Citadelle, Liège
- Canada (8):
  - Foothills Medical Centre, Calgary
  - Queen Elizabeth II Heath Sciences, Halifax
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal
  - Ottawa Heart Institute, Ottawa
  - Institut de Cardiologie de Quebec (Hospital Laval), Québec
  - Saint John Regional Hospital - New Brunswick Heart Centre, Saint John
  - Toronto General Hospital, Toronto
  - St. Paul's Hospital, Vancouver
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - CHRU Hopital de Pontchaillou, Rennes
  - CHU Rangueil Toulouse, Toulouse
  - Clinique Pasteur Toulouse, Toulouse
- Germany (14):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitatsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - Immanuelklinikum Bernau und Herzzentrum Brandenburg, Bernau
  - St Johannes Hospital, Dortmund
  - Herzzentrum Dresden GmbH Universitatsklinik, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universitat Frankfurt, Frankfurt
  - Universitatsmedizin Gottingen Georg-August-Universitat, Göttingen
  - Asklepios Klinikum St Georg, Hamburg
  - UKE Hamburg (Universitatsklinik Eppendorf), Hamburg
  - Universitatsklinikum Jena, Jena
  - Stadtisches Klinikum Karlsruhe gGmbH Medizinischen Klinik I, Karlsruhe
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum Munchen des Freistaates Bayern, München
- Kaplan Medical Center, Rehovot, Israel
- Italy (9):
  - Clinica Citta di Alessandria, Alessandria
  - Azienda Ospedali V. Emanuele Ferrarotto E S. Bambino, Catania
  - Fondazione Toscana Gabriele Monasterio - Ospedale del Cuore, Massa
  - Istituto Sant'Ambrogio, Milan
  - Ospedale Niguarda Ca'Granda, Milan
  - Ospedale San Raffaele, Milan
  - PoliclinicoSan Donato, Milan
  - Centro Cardiologico Monzino, Milan
  - Policlinico di Monza, Monza
- Vilnius University Hospital Santarisku KLinikos, Vilnius, Lithuania
- Netherlands (2):
  - OLVG, Amsterdam
  - Medisch Centrum Leeuwarden, Leeuwarden
- Spain (3):
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Clinico Universitario Virgen de Arrixaca, El Palmar
  - Hospital Universitario Virgen Macarena, Seville
- Universitatspital Spital Zurich, Zurich, Switzerland
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast
  - The Royal Sussex Country Hospital, Brighton
  - Kings College Hospital, London
  - Morriston hospital-ABM University Health Board, Morriston

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puri R, Thiele H, Fichtlscherer S, Westermann D, Makkar R, Waksman R, Hakmi S, Sondergaard L, Groh M, Montarello JK, Kempfert J, Yong G, Bedogni F, Maisano F, Worthley SG, Rodes-Cabau J, Fontana GP, Mollmann H. Five-Year Clinical Outcomes and Durability of a Self-Expanding Transcatheter Heart Valve With Intra-Annular Leaflets. Circ Cardiovasc Interv. 2025 Dec;18(12):e015430. doi: 10.1161/CIRCINTERVENTIONS.125.015430. Epub 2025 Oct 24. PMID 41133305
- [Derived] Sondergaard L, Rodes-Cabau J, Hans-Peter Linke A, Fichtlscherer S, Schafer U, Kuck KH, Kempfert J, Arzamendi D, Bedogni F, Asch FM, Worthley S, Maisano F. Transcatheter Aortic Valve Replacement With a Repositionable Self-Expanding Prosthesis: The PORTICO-I Trial 1-Year Outcomes. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2859-2867. doi: 10.1016/j.jacc.2018.09.014. Epub 2018 Sep 24. PMID 30261238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 973 subjects who were screened in Cohort A, 941 underwent an implant attempt with a Portico THV. Subjects in Cohort B were implanted in previous St. Jude Medical sponsored regulatory (pre-market) investigations and first-in-human trials, and consented for participation after completion of 1 year follow-up in their initial study.
Pre-assignment Details: The first subject was enrolled on April 16, 2013 and the last subject was enrolled on June 28, 2017. Among the 973 subjects who were screened initially in Cohort A, 32 were excluded due to screen failures or exit without a Portico implant attempt. Hence only 941 subjects from Cohort A and 59 from Cohort B were considered for baseline, endpoint and safety analyses.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 941 | 59
Completed | 398 | 34
Not Completed | 543 | 25
Not completed — Withdrawal by Subject | 102 | 5
Not completed — Death | 382 | 18
Not completed — Lost to Follow-up | 31 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Patient Non-Compliance | 1 | 0
Not completed — Study Stopped/Terminated at Site | 5 | 0
Not completed — Other Reasons | 19 | 0

BASELINE CHARACTERISTICS:
Population: Of the 973 subjects who were screened in Cohort A, 32 subjects did not undergo an implant attempt with Portico THV. Hence only 941 subjects from Cohort A and 59 from Cohort B were considered for baseline, endpoint and safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 941 | 59 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.4 (5.9) | 82.3 (4.6) | 82.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 618 | 37 | 655
  Male | 323 | 22 | 345
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 22 | 0 | 22
  Switzerland | 4 | 0 | 4
  Spain | 35 | 0 | 35
  Canada | 60 | 0 | 60
  Netherlands | 29 | 12 | 41
  Belgium | 34 | 0 | 34
  Denmark | 56 | 1 | 57
  Italy | 133 | 0 | 133
  Israel | 2 | 0 | 2
  Australia | 129 | 7 | 136
  France | 20 | 0 | 20
  Lithuania | 7 | 0 | 7
  Germany | 410 | 39 | 449
NYHA Classification [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  Participants
    NYHA I: number analyzed (Participants) | 937 | 59 | 996
    NYHA I | 29 | 0 | 29
    NYHA II: number analyzed (Participants) | 937 | 59 | 996
    NYHA II | 309 | 16 | 325
    NYHA III: number analyzed (Participants) | 937 | 59 | 996
    NYHA III | 554 | 41 | 595
    NYHA IV: number analyzed (Participants) | 937 | 59 | 996
    NYHA IV | 45 | 2 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With All-cause Mortality
Description: Percentage of participants that died for any reason at 1 year post implantation
Time Frame: 1 year post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants | 12.1 [10.1 to 14.4]

2. Secondary Outcome: Percentage of Participants With All Cause Mortality in Cohort A
Description: Percentage of participants that died for any reason at 30 days through 5 years post implantation
Time Frame: 30 days through 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  30 days | 2.7
  1 year | 12.0
  2 years | 19.5
  3 years | 27.0
  4 years | 35.7
  5 years | 44.3

3. Secondary Outcome: Number of Participants With All-cause Mortality (30 Days, Annually From 1 Year Through 5 Years) in Cohort B
Description: Number of participants who died for any reason at different time points such as 30 days, 1 year, 2 years, 3 years, 4 years and 5 years.
Time Frame: 30 days through 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  2 years | 4
  3 years | 4
  4 years | 5
  5 years | 5

4. Secondary Outcome: Percentage of Participants With Cardiovascular Mortality as Defined by the Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants that died for cardiovascular or unknown reasons as defined by VARC-2 at 30 days through 5 years post implantation
Time Frame: 30 days through 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  30 days | 2.5
  1 year | 6.6
  2 year | 9.8
  3 year | 13.1
  4 year | 18.5
  5 year | 24.1

5. Secondary Outcome: Number of Participants With Cardiovascular Mortality Occurring at Each Time Window (30 Days, 1 Year, 2 Years, 3 Years, 4 Years and 5 Years) in Cohort B
Description: as for outcome 3
Time Frame: 30 days through 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  2 years | 0
  3 years | 4
  4 years | 2
  5 years | 4

6. Secondary Outcome: Percentage of Participants With Non-Cardiovascular Mortality as Defined by the Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants that died for any reason at 30 days through 5 years post implantation
Time Frame: 30 days through 5 years post implant
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  30 days | 0.2
  1 year | 5.8
  2 years | 10.8
  3 years | 16.0
  4 years | 21.1
  5 years | 26.6

7. Secondary Outcome: Number of Participants With Non-Cardiovascular Mortality Occurring at Each Time Window (30 Days, 1 Year, 2 Years, 3 Years, 4 Years and 5 Years) in Cohort B
Description: as for outcome 3
Time Frame: 30 days through 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  2 years | 1
  3 years | 3
  4 years | 2
  5 years | 1

8. Secondary Outcome: Percentage of Participants With Myocardial Infarction as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a myocardial infarction as defined by VARC-2 at 30 days through 5 years post implantation post implantation
Time Frame: 30 days through 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  30 days | 1.6
  1 year | 2.5
  2 years | 3.2
  3 years | 3.6
  4 years | 4.9
  5 years | 6.5

9. Secondary Outcome: Number of Participants With Myocardial Infarction as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a myocardial infarction as defined by VARC-2 at 30 days through 5 years post implantation post implantation
Time Frame: 30 days through 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  2 years | 0
  3 years | 1
  4 years | 1
  5 years | 0

10. Secondary Outcome: Percentage of Participants With Vascular Access Site Complication as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with vascular access site complication (major or minor) as defined by VARC-2 at 30 days post implantation
Time Frame: 30 days post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Major | 7.0
  Minor | 6.2

11. Secondary Outcome: Percentage of Participants With Bleeding Events as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a bleeding events (life threatening, major or minor) as defined by VARC-2 at 30 days post implantation
Time Frame: 30 days post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Life threatening | 3.3
  Major | 8.3
  Minor | 8.9

12. Secondary Outcome: Percentage of Participants With Stage 1, 2 and 3 Acute Kidney Injury as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a Stage 1, 2 or Stage 3 acute kidney injury as defined by VARC-2 at 30 days post implantation
Time Frame: 30 days post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Stage 1 | 0.4
  Stage 2 | 1.0
  Stage 3 | 2.0

13. Secondary Outcome: Mean Prosthetic Valve Function as Defined by Valve Academic Research Consortium-2 (VARC-2) (Aortic Valve Area)
Description: The aortic valve area as interpreted by an independent echocardiographic core laboratory at 30 days through 5 years post implantation
Time Frame: 30 days through 5 years post implant
Population: The data for the number of participants available at the time has been provided. For Cohort A, a total of 941 subjects participated in the study; however, only 574 were available for AVA analysis.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 574 | 59
cm^2
  30 days | 1.78 (0.48) | NA (NA) — Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
  1 year: number analyzed (Participants) | 476 | 59
  1 year | 1.74 (0.48) | NA (NA) — Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
  2 years: number analyzed (Participants) | 302 | 36
  2 years | 1.84 (0.57) | 1.88 (0.49)
  3 years: number analyzed (Participants) | 166 | 23
  3 years | 1.76 (0.53) | 1.76 (0.45)
  4 years: number analyzed (Participants) | 211 | 19
  4 years | 1.76 (0.57) | 1.88 (0.48)
  5 years: number analyzed (Participants) | 123 | 16
  5 years | 1.84 (0.47) | 1.74 (0.48)

14. Secondary Outcome: Mean Prosthetic Valve Function as Defined by Valve Academic Research Consortium-2 (VARC-2) (Mean Transvalvular Gradient)
Description: The mean transvalvular gradient as interpreted by an independent echocardiographic core laboratory at 30 days through 5 years post implantation
Time Frame: 30 days through 5 years post implant
Population: The data for the number of participants available at the time has been provided. For Cohort A, a total of 941 subjects participated in the study; however, only 684 were available for mean aortic gradient analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 684 | 59
mmHg
  30 days | 8.58 (3.89) | NA (NA) — Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
  1 year: number analyzed (Participants) | 570 | 59
  1 year | 8.67 (4.11) | NA (NA) — Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
  2 years: number analyzed (Participants) | 365 | 45
  2 years | 7.81 (3.78) | 8.04 (3.00)
  3 years: number analyzed (Participants) | 237 | 34
  3 years | 7.61 (4.29) | 7.34 (4.03)
  4 years: number analyzed (Participants) | 285 | 31
  4 years | 7.99 (4.10) | 7.69 (4.07)
  5 years: number analyzed (Participants) | 181 | 23
  5 years | 6.69 (3.52) | 6.44 (4.00)

15. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Classification of Heart Failure
Description: The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity:
  Class I - No symptoms and no limitation in ordinary physical activity; Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity; Class III - Marked limitation in activity due to symptoms; Class IV - Severe limitations.
Time Frame: 30 days post implant
Population: The data for the number of participants available at the time has been provided
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 808 | 54
Participants
  Class I | 298 | 13
  Class II | 405 | 35
  Class III | 98 | 6
  Class IV | 7 | 0

16. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Classification of Heart Failure
Description: as for outcome 15
Time Frame: 1 year post implant
Population: The data for the number of participants available at the time has been provided
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 699 | 59
Participants
  Class I | 289 | 23
  Class II | 356 | 25
  Class III | 51 | 10
  Class IV | 3 | 1

17. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Classification of Heart Failure
Description: as for outcome 15
Time Frame: 2 years post implant
Population: The data for the number of participants available at the time has been provided
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 595 | 46
Participants
  Class I | 244 | 14
  Class II | 283 | 22
  Class III | 64 | 10
  Class IV | 4 | 0

18. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Classification of Heart Failure
Description: as for outcome 15
Time Frame: 3 years post implant
Population: The data for the number of participants available at the time has been provided
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 509 | 44
Participants
  Class I | 194 | 15
  Class II | 251 | 19
  Class III | 62 | 9
  Class IV | 2 | 1

19. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Classification of Heart Failure
Description: as for outcome 15
Time Frame: 4 years post implant
Population: The data for the number of participants available at the time has been provided
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 423 | 39
Participants
  Class I | 147 | 7
  Class II | 211 | 26
  Class III | 59 | 5
  Class IV | 6 | 1

20. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Classification of Heart Failure
Description: as for outcome 15
Time Frame: 5 years post implant
Population: The data for the number of participants available at the time has been provided
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 345 | 34
Participants
  Class I | 113 | 11
  Class II | 174 | 14
  Class III | 54 | 8
  Class IV | 4 | 1

21. Secondary Outcome: Mean Six Minute Walk Test (6MWT)
Description: Distance in metres that the participant can walk in 6 minutes. The six-minute walking test (6MWT) is a commonly used objective measure of functional exercise capacity in individuals with moderately severe impairment.
Time Frame: 30 days through 5 years post implant
Population: The data for the number of participants available at the time has been provided. For Cohort A, a total of 941 subjects participated in the study; however, only 569 were available for 6 minute walk test.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 569 | 59
meter
  30 days: number analyzed (Participants) | 569 | 46
  30 days | 276.3 (117.5) | 250.60 (104.61)
  1 year: number analyzed (Participants) | 495 | 50
  1 year | 285.75 (112.12) | 257.18 (97.96)
  2 years: number analyzed (Participants) | 319 | 35
  2 years | 276.4 (116.2) | 253.4 (119.8)
  3 years: number analyzed (Participants) | 176 | 28
  3 years | 283.4 (119.4) | 244.4 (111.6)
  4 years: number analyzed (Participants) | 145 | 23
  4 years | 288.4 (106.2) | 236.4 (100.0)
  5 years: number analyzed (Participants) | 121 | 15
  5 years | 286.4 (110.9) | 197.5 (107.7)

22. Secondary Outcome: Mean Quality of Life Assessment in Cohort A
Description: EuroQuol-5 Dimensions (EQ5D) is a standardized instrument for use as a measure of health outcome applicable to a wide range of health conditions and treatments. A visual analog scale (VAS) for health is also included in the measure as a patient-reported estimate of overall health status. This scale ranges between 0-100, where 0 is 'the worst health you can imagine' and 100 is 'the best health you can imagine'.
Time Frame: 30 days and 1 year post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up. For Cohort A, a total of 941 subjects participated in the study; however, only 774 were available for EQ5D analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A
Number analyzed (Participants) | 774
score on a scale
  30 days | 67.3 (18.0)
  1 year: number analyzed (Participants) | 670
  1 year | 68.8 (17.7)

23. Secondary Outcome: Percentage of Participants With Transient Ischemic Attack in Cohort A
Description: Percentage of participants with transient ischemic attack as defined by VARC-2 at 30 days through 5 years post implantation
Time Frame: 30 days through 5 years post implantation
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  30 days | 0.4
  1 year | 1.4
  2 years | 1.9
  3 years | 1.9
  4 years | 2.5
  5 years | 2.8

24. Secondary Outcome: Number of Participants With Transient Ischemic Attack in Cohort B
Description: Number of participants with transient ischemic attack as defined by VARC-2 at 30 days through 5 years post implantation
Time Frame: 30 days through 5 years post implantation
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  2 years | 1
  3 years | 0
  4 years | 0
  5 years | 0

25. Secondary Outcome: Percentage of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 30 days post implantation
Time Frame: 30 days post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Disabling | 1.4
  Non-disabling | 1.2

26. Secondary Outcome: Percentage of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 1 year post implantation
Time Frame: 1 year post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Disabling | 2.1
  Non-disabling | 2.0

27. Secondary Outcome: Percentage of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 2 years post implantation
Time Frame: 2 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Disabling | 3.2
  Non-disabling | 3.2

28. Secondary Outcome: Percentage of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 3 years post implantation
Time Frame: 3 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Disabling | 4.3
  Non-disabling | 3.9

29. Secondary Outcome: Percentage of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 4 years post implantation
Time Frame: 4 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Disabling | 6.3
  Non-disabling | 4.3

30. Secondary Outcome: Percentage of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 5 years post implantation
Time Frame: 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  Disabling | 7.8
  Non-disabling | 4.7

31. Secondary Outcome: Number of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 2 years post implantation
Time Frame: 2 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  Disabling | 0
  Non-disabling | 0

32. Secondary Outcome: Number of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 3 years post implantation
Time Frame: 3 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  Disabling | 0
  Non-disabling | 0

33. Secondary Outcome: Number of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 4 years post implantation
Time Frame: 4 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  Disabling | 0
  Non-disabling | 0

34. Secondary Outcome: Number of Participants With Stroke as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a stroke (disabling and non-disabling) as defined by VARC-2 at 5 years post implantation
Time Frame: 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  Disabling | 0
  Non-disabling | 0

35. Secondary Outcome: Percentage of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 30 days post implantation
Time Frame: 30 days post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  New-onset atrial fibrillation | 4.0
  New pacemaker implant in pacemaker naïve patients | 19.0
  Overall PM implantation | 17.3

36. Secondary Outcome: Percentage of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 1 year post implantation
Time Frame: 1 year post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  New-onset atrial fibrillation | 5.3
  New pacemaker implant in pacemaker naïve patients | 21.2
  Overall PM implantation | 19.4

37. Secondary Outcome: Percentage of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 2 years post implantation
Time Frame: 2 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  New-onset atrial fibrillation | 5.9
  New pacemaker implant in pacemaker naïve patients | 22.4
  Overall PM implantation | 20.4

38. Secondary Outcome: Percentage of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 3 years post implantation
Time Frame: 3 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  New-onset atrial fibrillation | 7.3
  New pacemaker implant in pacemaker naïve patients | 23.6
  Overall PM implantation | 21.6

39. Secondary Outcome: Percentage of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 4 years post implantation
Time Frame: 4 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  New-onset atrial fibrillation | 8.8
  New pacemaker implant in pacemaker naïve patients | 25.4
  Overall PM implantation | 23.2

40. Secondary Outcome: Percentage of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort A
Description: Percentage of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 5 years post implantation
Time Frame: 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 941
percentage of participants
  New-onset atrial fibrillation | 9.5
  New pacemaker implant in pacemaker naïve patients | 27.7
  Overall PM implantation | 25.3

41. Secondary Outcome: Number of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 2 years post implantation
Time Frame: 2 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  New-onset atrial fibrillation | 1
  New pacemaker implant in pacemaker naïve patients | 1
  Overall PM implantation | 1

42. Secondary Outcome: Number of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 3 years post implantation
Time Frame: 3 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  New-onset atrial fibrillation | 0
  New pacemaker implant in pacemaker naïve patients | 0
  Overall PM implantation | 0

43. Secondary Outcome: Number of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 4 years post implantation
Time Frame: 4 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  New-onset atrial fibrillation | 2
  New pacemaker implant in pacemaker naïve patients | 0
  Overall PM implantation | 0

44. Secondary Outcome: Number of Participants With Conduction Disturbances and Cardiac Arrythmias as Defined by Valve Academic Research Consortium-2 (VARC-2) in Cohort B
Description: Number of participants with a conduction disturbances and cardiac arrhythmias as defined by VARC-2 at 5 years post implantation
Time Frame: 5 years post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 59
Participants
  New-onset atrial fibrillation | 1
  New pacemaker implant in pacemaker naïve patients | 0
  Overall PM implantation | 0

45. Secondary Outcome: Percentage of Participants With Prosthetic Valve Function as Defined by Valve Academic Research Consortium-2 (VARC-2) (Paravalvular Aortic Regurgitation) in Cohort A
Description: Percentage of participants with a paravalvular aortic regurgitation as defined by VARC-2 at 30 days post implantation
Time Frame: 30 days post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 689
percentage of participants
  None/trace/trivial | 28.4
  Mild | 67.6
  Moderate | 3.9
  Severe | 0.0

46. Secondary Outcome: Percentage of Participants With Prosthetic Valve Function as Defined by Valve Academic Research Consortium-2 (VARC-2) (Paravalvular Aortic Regurgitation) in Cohort A
Description: Percentage of participants with a paravalvular aortic regurgitation as defined by VARC-2 at 1 year post implantation
Time Frame: 1 year post implant
Population: Cohort B subjects in the Portico I study scheduled follow-up visit starting with the 2 year follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 575
percentage of participants
  None/trace/trivial | 29.7
  Mild | 67.7
  Moderate | 2.6
  Severe | 0.0

47. Secondary Outcome: Percentage of Participants With Prosthetic Valve Function as Defined by Valve Academic Research Consortium-2 (VARC-2) (Paravalvular Aortic Regurgitation)
Description: Percentage of participants with a paravalvular aortic regurgitation as defined by VARC-2 at 2 years post implantation
Time Frame: 2 years post implant
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 344 | 40
percentage of participants
  None/trace/trivial | 56.1 | 57.5
  Mild | 42.4 | 42.5
  Moderate | 1.5 | 0.0
  Severe | 0.0 | 0.0

48. Secondary Outcome: Percentage of Participants With Prosthetic Valve Function as Defined by Valve Academic Research Consortium-2 (VARC-2) (Paravalvular Aortic Regurgitation)
Description: Percentage of participants with a paravalvular aortic regurgitation as defined by VARC-2 at 3 years post implantation
Time Frame: 3 years post implant
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 248 | 34
percentage of participants
  None/trace/trivial | 64.9 | 70.6
  Mild | 34.7 | 29.4
  Moderate | 0.4 | 0.0
  Severe | 0.0 | 0.0

49. Secondary Outcome: Percentage of Participants With Prosthetic Valve Function as Defined by Valve Academic Research Consortium-2 (VARC-2) (Paravalvular Aortic Regurgitation)
Description: Percentage of participants with a paravalvular aortic regurgitation as defined by VARC-2 at 4 years post implantation
Time Frame: 4 years post implant
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 188 | 28
percentage of participants
  None/trace/trivial | 53.2 | 50.0
  Mild | 45.7 | 50.0
  Moderate | 1.1 | 0.0
  Severe | 0.0 | 0.0

50. Secondary Outcome: Percentage of Participants With Prosthetic Valve Function as Defined by Valve Academic Research Consortium-2 (VARC-2) (Paravalvular Aortic Regurgitation)
Description: Percentage of participants with a paravalvular aortic regurgitation as defined by VARC-2 at 5 years post implantation
Time Frame: 5 years post implant
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 182 | 23
percentage of participants
  None/trace/trivial | 69.8 | 69.6
  Mild | 28.6 | 30.4
  Moderate | 1.6 | 0.0
  Severe | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: 5 Year
Description: The 5-year KM rate of all-cause mortality is estimated on exact 1826 days post procedure, so 366 are the # of death happened before this time.
  In the withdrawal table, the # of death, 382, are counted based on visit window of the 5 years visit. If a subject missed 5 years visit and the death happened before the upper window of 5 years visit, the death will be counted. So normally the withdrawal table will show more death than the KM rate table.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 382/941 | 18/59
Serious Adverse Events (participants affected / at risk) | 754/941 | 40/59
Other Adverse Events (participants affected / at risk) | 526/941 | 22/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=941) | Cohort B (N=59)
Clinical significant bleeding (Blood and lymphatic system disorders) | 67 | 3
Life threatening bleeding (Blood and lymphatic system disorders) | 31 | 0
Major bleeding (Blood and lymphatic system disorders) | 74 | 0
Minor bleeding (Blood and lymphatic system disorders) | 15 | 0
Not clinical significant bleeding (Blood and lymphatic system disorders) | 17 | 1
Arrhythmia / Conduction abnormality (Cardiac disorders) | 256 | 3
Coronary obstruction (Cardiac disorders) | 1 | 0
Endocarditis (Cardiac disorders) | 7 | 0
New Onset of Atrial Fibrillation (Cardiac disorders) | 25 | 1
Peri-Procedural MI (Cardiac disorders) | 11 | 0
Prosthetic aortic valve regurgitation (Cardiac disorders) | 7 | 0
Prosthetic aortic valve stenosis (Cardiac disorders) | 2 | 0
Spontaneous MI (Cardiac disorders) | 34 | 2
Disabling stroke (General disorders) | 53 | 0
Non-Disabling stroke (General disorders) | 35 | 0
Other (General disorders) | 597 | 33
TIA (General disorders) | 17 | 1
Stage 1 AKI (Renal and urinary disorders) | 6 | 0
Stage 2 AKI (Renal and urinary disorders) | 8 | 0
Stage 3 AKI (Renal and urinary disorders) | 39 | 0
Undetermined AKI (Renal and urinary disorders) | 13 | 2
Need for second TAVI (Surgical and medical procedures) | 8 | 0
Pacemaker implantation (Surgical and medical procedures) | 204 | 1
Major vascular complications (Vascular disorders) | 65 | 0
Minor vascular complications (Vascular disorders) | 14 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=941) | Cohort B (N=59)
Clinical significant bleeding (Blood and lymphatic system disorders) | 3 | 0
Life threatening bleeding (Blood and lymphatic system disorders) | 1 | 0
Major bleeding (Blood and lymphatic system disorders) | 5 | 0
Minor bleeding (Blood and lymphatic system disorders) | 69 | 0
Not clinical significant bleeding (Blood and lymphatic system disorders) | 7 | 0
Endocarditis (Cardiac disorders) | 3 | 0
New Onset of Atrial Fibrillation (Cardiac disorders) | 50 | 3
Peri-Procedural MI (Cardiac disorders) | 2 | 0
Prosthetic aortic valve regurgitation (Cardiac disorders) | 27 | 0
Prosthetic aortic valve stenosis (Cardiac disorders) | 6 | 0
Arrhythmia / Conduction abnormality (Cardiac disorders) | 284 | 5
Other (General disorders) | 312 | 17
TIA (General disorders) | 5 | 0
Stage 1 AKI (Renal and urinary disorders) | 3 | 0
Stage 2 AKI (Renal and urinary disorders) | 2 | 1
Stage 3 AKI (Renal and urinary disorders) | 2 | 0
Undetermined AKI (Renal and urinary disorders) | 5 | 0
Need for second TAVI (Surgical and medical procedures) | 5 | 0
Pacemaker implantation (Surgical and medical procedures) | 8 | 0
Major vascular complications (Vascular disorders) | 2 | 0
Minor vascular complications (Vascular disorders) | 45 | 0
Undetermined vascular complications (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Cohort B entered the study after completion of their 1 year follow-up in other trials, therefore there are no results for Cohort B prior to 2 years collected in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT01802788/Prot_SAP_000.pdf